CLINICAL TRIAL: NCT05550402
Title: Comparison of Parasympathetic Activity in Mild, Moderate, and Severe Asthma With Fixed Airway Obstruction
Brief Title: Role of Parasympathetic Activity in Mild to Severe Asthma With Fixed Airway Obstruction (PARASMA Study)
Acronym: PARASMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Narongwit Nakwan, Asst. Prof., Hat Yai Medical Education Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 454554
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Airway Obstruction; Airway Remodeling; Parasympathetic Nervous System Diseases
Keywords: asthma; fixed airway obstruction; spirometry; parasympathetic activity; well controlled
MeSH Terms: conditions — Asthma; Airway Obstruction; Airway Remodeling; Autonomic Nervous System Diseases | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Salbutamol then ipratropium (Active Comparator): Visit 1, After predosed spirometry is done, the patients will be received 4 puffs of salbutamol. 30 minutes later, if they meet the criteria of fixed airway obstruction based on ATS criteria, then they will continue to undergo serial spirometry at 1, 2, 3, and 4 hours. Then, the patients requested to be administered 4 puffs of ipratropium and do spirometry at 4.5 and 5 hours.
  Interventions: Drug: Salbutamol; Drug: Ipratropium Bromide
- Ipratropium then salbutamol (Active Comparator): Visit 2, After predosed spirometry is done, the patients will be received 4 puffs of ipratropium they will continue to undergo serial spirometry at 30 minutes,1, 2, 3, and 4 hours. Then, the patients requested to be administered 4 puffs of salbutamol and do spirometry at 4.5 and 5 hours.
  Interventions: Drug: Salbutamol; Drug: Ipratropium Bromide
- Salbutamol plus ipratropium (Active Comparator): Visit 3, After predosed spirometry is done, the patients will be received 4 puffs of a placebo, and they will do spirometry at 30 minutes, 1 and 2 hours (Placebo arm). Then, the patients requested to be administered 4 puffs of ipratropium and 4 puffs of salbutamol and do spirometry at 4.5 and 5 hours (Salbutamol plus ipratropium)
  Interventions: Drug: Salbutamol plus Ipratropium Bromide
- Placebo (Placebo Comparator): Visit 3, After predosed spirometry is done, the patients will be received 4 puffs of a placebo, and they will do spirometry at 30 minutes, 1 and 2 hours (Placebo arm).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Salbutamol — Visit 1, After predosed spirometry is done, the patients will be received 4 puffs of salbutamol. 30 minutes later, if they meet the criteria of fixed airway obstruction based on ATS criteria, then they will continue to undergo serial spirometry at 1, 2, 3, and 4 hours. Then, the patients requested to be administered 4 puffs of ipratropium and do spirometry at 4.5 and 5 hours.
  Other Names: ventolin
  Arms: Ipratropium then salbutamol; Salbutamol then ipratropium
Drug: Ipratropium Bromide — Visit 2, After predosed spirometry is done, the patients will be received 4 puffs of ipratropium they will continue to undergo serial spirometry at 30 minutes,1, 2, 3, and 4 hours. Then, the patients requested to be administered 4 puffs of salbutamol and do spirometry at 4.5 and 5 hours.
  Other Names: Atrovent
  Arms: Ipratropium then salbutamol; Salbutamol then ipratropium
Drug: Salbutamol plus Ipratropium Bromide — Visit 3, After predosed spirometry is done, the patients will be received 4 puffs of a placebo, and they will do spirometry at 30 minutes, 1 and 2 hours (Placebo arm). Then, the patients requested to be administered 4 puffs of ipratropium and 4 puffs of salbutamol and do spirometry at 4.5 and 5 hours (Salbutamol plus ipratropium arm)
  Arms: Salbutamol plus ipratropium
Other: Placebo — Visit 3, After predosed spirometry is done, the patients will be received 4 puffs of a placebo, and they will do spirometry at 30 minutes, 1 and 2 hours (Placebo arm).
  Arms: Placebo

SUMMARY:
In asthma, the significant role of pathogenesis is chronic airway inflammation, bronchial hyperresponsiveness, and variable airflow obstruction. Asthma with irreversible or fixed airflow obstruction (FAO) is a clinical phenotype resulting from chronic airway inflammation with having longer disease duration, suggesting that airway remodeling contributes to the decline in lung function seen in individuals with asthma. Although this condition frequently occurs in patients with severe asthma, there are pieces of evidence occurring in those with mild to moderate asthma. According to previous research, low lung function, FEV1 less than 60% predicted, is a robust independent predictor of subsequent asthma attacks and other asthma outcomes, including asthma control and SABA use. In a recent study, the patients with mild to moderate asthma who received mild to medium dosed inhaled corticosteroid plus long-acting beta-2 agonist with or without asthma control showed evidence of FAO with or without bronchodilator reversibility. Therefore parasympathetic activity may be affected by FAO in those patients. The autonomic nervous system plays an essential role in asthma, especially from the parasympathetic, promoting bronchoconstriction and regulating airway inflammation and remodeling. This study hypothesizes that a cholinergic mechanism may play a significant role in FAO across patients with mild, moderate, and severe asthma. This might increase the fundamental evidence leading to early-step treatment with anti-cholinergic medication in early asthma severity driven by FAO.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients classified by severity Mild (achieved control with using low-dose ICS or as-needed ICS-formoterol) or Moderate (achieved controlled with using low-dose ICS/LABA or Severe ((achieved controlled with using medium to high dose ICS/LABA)
* Post-bronchodilator (Salbutamol) FEV1/FVC ratio less than 0.75 or below the Lower Limit of Normal (LLN) and Post-bronchodilator (Salbutamol) FEV1 predicted < 80% with or without bronchodilator response
* History of smoking less than 10 pack-years or current smoking
* Patients who able to do spirometry without contraindication
* asthma control was defined by ACQ6 < 1.5

Exclusion Criteria:

* Contraindication for spirometry
* Chest x-ray suggested any chronic lung diseased
* Contraindication for anticholinergic drug
* History of asthma exacerbation within 12 weeks before visit 1
* History of taking LAMA within 6 months before visit 1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Average FEV1 | 6 hour
  FEV1 determined from serial spirometry and calculated on the basis of area under the curve

SECONDARY OUTCOMES:
FEV1 at 6 h | 6 hour
  FEV1 at 6 hours post-dose
Maximum FEV1 | 6 hour
  Maximum FEV1 over the 6-hour serial assessments

CONTACTS AND LOCATIONS:
Overall Officials: Narongwit Nakwan, M.D., Principal Investigator — Hatyai medical Education Center, Hatyai Hospital
Locations (1):
- Hatyai Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided